CLINICAL TRIAL: NCT03587272
Title: Minimizing Toxicity in HLA-identical Sibling Donor Transplantation for Children With Sickle Cell Disease
Acronym: SUN
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Robert Nickel (Other)
Collaborators: Alberta Children's Hospital (Other); The Hospital for Sick Children (Other); Levine Children's Hospital (Other); Ann & Robert H Lurie Children's Hospital of Chicago (Other); Nationwide Children's Hospital (Other); The Children's Hospital at Montefiore (Other); Columbia University (Other)
Responsible Party: Sponsor-Investigator, Robert Nickel, Principal Investigator, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB 10322
Record Dates: First submitted 2018-06-06; First posted 2018-07-16 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Alemtuzumab; Whole-Body Irradiation; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SUN regimen (Experimental): Alemtuzumab, low dose total body irradiation, Sirolimus
  HLA-identical sibling donor transplantation using alemtuzumab, low dose total-body irradiation, and sirolimus (Sickle transplant Using a Nonmyeloablative approach, "SUN") can decrease the toxicity of transplant while achieving a high cure rate for children with sickle cell disease (SCD).
  Interventions: Drug: Alemtuzumab, low dose total body irradiation, Sirolimus

INTERVENTIONS:
Drug: Alemtuzumab, low dose total body irradiation, Sirolimus — The conditioning regimen (SUN regimen) will consist of alemtuzumab daily for 5 days (total dose 1 mg/kg) and low dose total body irradiation (TBI) 300 cGY on Day -2 with gonadal shielding if possible. The HSCT graft will be G-CSF mobilized PBSCs with minimum CD34+ of 5 x106/kg recipient weight, goal of 10 x 106/kg (no upper limit). A peripheral blood stem cell (PBSC) graft was selected as it engrafts faster than bone marrow and would lead to shorter period of neutropenia and infection and less thrombocytopenia and need for platelet transfusion.
  GVHD prophylaxis will be sirolimus with a loading dose 3 mg/m2 on day -1. Sirolimus will be continued at 1 mg/m2/day starting on day 0 and dose adjusted to maintain a target trough level 5-15 ng/mL for the first 3 months and 5-10 ng/mL for the remainder of the first year.

SUMMARY:
This multisite prospective study seeks to determine if HLA-identical sibling donor transplantation using alemtuzumab, low dose total-body irradiation, and sirolimus (Sickle transplant Using a Nonmyeloablative approach, "SUN") can decrease the toxicity of transplant while achieving a high cure rate for children with sickle cell disease (SCD).

DETAILED DESCRIPTION:
This is a prospective, multicenter phase II study of HLA-identical sibling donor HSCT in 30 pediatric patients with SCD using nonmyeloablative conditioning with alemtuzumab, total-body irradiation, and sirolimus. The primary Objective of this study is to determine if the SUN regimen can decrease the incidence of grade II-IV acute graft-versus host disease (GVHD) by day +100 while maintaining similar disease-free survival compared to establish HLA-identical donor hematopoietic stem cell transplant (HSCT) regimens in children with SCD. The secondary Objective is to determine if health-related quality of life (HRQoL) for children undergoing SUN HSCT is preserved during the early post-transplant time period. To determine if the SUN regimen can decrease the number of platelet transfusions compared to established HLA-identical HSCT regimens in children with SCD. The tertiary/Exploratory Objectives: To describe other markers of toxicity (duration of neutropenia, mucositis, length of hospitalization) and indicators of a successful HSCT (HRQoL at 1 year, proportion needing additional immunosuppression during the first year, proportion able to wean sirolimus at 1 year).

With protocol version 5.0, added new secondary objective to determine if the change from intravenous to subcutaneous alemtuzumab and the addition of post-HSCT G-CSF can decrease the incidence of poor donor engraftment.

ELIGIBILITY:
Inclusion criteria:

Patients with genotypes hemoglobin SS and Sβ0 thalassemia must have at least one of the following:

* History of an abnormal transcranial Doppler measurement defined as TCD velocity ≥200 cm/sec by the non-imaging technique (or ≥185 cm/sec by the imaging technique) measured at a minimum of two separate occasions.
* History of cerebral infarction on brain MRI (overt stroke, or silent stroke if ≥3 mm in one dimension, visible in two planes on fluid-attenuated inversion recovery T2-weighted images).
* History of two or more episodes of acute chest syndrome (ACS) in lifetime.
* History of three or more SCD pain events requiring treatment with an opiate or IV pain medication (inpatient or outpatient) in lifetime.
* History of any hospitalization for SCD pain or ACS while receiving hydroxyurea treatment.
* History of two or more episodes of priapism (erection lasting ≥4 hours or requiring emergent medical care).
* Administration of regular RBC transfusions (≥8 transfusions in the previous 12 months).
* At least two episodes of splenic sequestration requiring red blood cell transfusion or splenectomy after at least one episode of splenic sequestration.

Patients with all other sickle genotypes (hemoglobin SC, Sβ+ thalassemia) must have at least one of the following:

* Clinically significant neurologic event (overt stroke).
* History of two or more episodes of ACS in the 2-years period preceding enrollment.
* History of three or more SCD pain events requiring treatment with an opiate or IV pain medication (inpatient or outpatient) in the 1-year period preceding enrollment.
* History of any hospitalization for SCD pain or ACS while receiving hydroxyurea treatment.
* History of two or more episodes of priapism (erection lasting ≥4 hours or requiring emergent medical care).
* Administration of regular RBC transfusions (≥8 transfusions in the previous 12 months).
* At least two episodes of splenic sequestration requiring red blood cell transfusion or splenectomy after at least one episode of splenic sequestration.

Exclusion Criteria:

* General: Life expectancy less than 6 months. Pregnant or breastfeeding patients.
* Infection Disease: Uncontrolled bacterial, viral or fungal infections (undergoing appropriate treatment and with progression of clinical symptoms) within 1 month prior to conditioning. Patients with febrile illness or suspected minor infection should await clinical resolution prior to starting conditioning. Patients with confirmed seropositivity for HIV and patients with active Hepatitis B or C determined by serology and/or NAAT are excluded.
* Liver: Direct (conjugated) bilirubin > 1.5 mg/dL, transaminases >5x upper limit of normal for age.
* Cardiac: Left ventricular shortening fraction <25% or ejection fraction <50% by ECHO.
* Kidney: Estimated creatinine clearance less than 60 mL/min/1.73m2.
* Pulmonary function: Diffusion capacity of carbon monoxide (DLCO) <35% (adjusted for hemoglobin). Baseline oxygen saturation <85% or PaO2 <70.
* Heme: History of RBC alloantibodies against donor RBC antigens (even if current antibody screen is negative). Major ABO incompatibility with donor.

Ages: 2 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-04-17 (Actual); Primary Completion 2030-11 (Estimated); Study Completion 2030-11 (Estimated)

PRIMARY OUTCOMES:
Acute GVHD | 100 days post transplant
  Acute grade II-IV GVHD

SECONDARY OUTCOMES:
PedsQL 4.0 Measurement model for the Pediatric Quality of Life Inventory | Day +30, and day +100 post transplant
  PedsQL 4.0 assessments of health related quality of life before/after transplant
Poor donor engraftment | day +365
  graft rejection, stem cell boost, or 1-year donor myeloid chimerism <50%

OTHER OUTCOMES:
Patient-Reported Outcomes Measurement Information System (PROMIS) | Day +30, and day +100 post transplant
  PROMIS assessments of health related quality of life before/after transplant
Platelet transfusion | 100 days post transplant
  Number of platelet transfusions

CONTACTS AND LOCATIONS:
Overall Officials: Robert Nickel, MD, Principal Investigator — Children's National Research Institute
Locations (7):
- United States (5):
  - Children's National Health System, Washington D.C., District of Columbia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Columbia University, New York, New York
  - Levine Children's Hospital, Charlotte, North Carolina
  - Nationwide Children's Hospital, Columbus, Ohio
- Canada (2):
  - Alberta Children's Hospital, Calgary, Alberta
  - The Hospital for Sick Children, Toronto, Ontario

REFERENCES:
- [Derived] Leonard A, Furstenau D, Abraham A, Darbari DS, Nickel RS, Limerick E, Fitzhugh C, Hsieh M, Tisdale JF. Reduction in vaso-occlusive events following stem cell transplantation in patients with sickle cell disease. Blood Adv. 2023 Jan 24;7(2):227-234. doi: 10.1182/bloodadvances.2022008137. PMID 36240296